CLINICAL TRIAL: NCT06288698
Title: Analyzing Enrolment and Engagement Trends in Individuals Confronting TBI: Insights From TBI Clinical Trials
Brief Title: Understanding Patient Engagement Trends in TBI Clinical Research
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 53955721
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: TBI
Keywords: TBI

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical trials, specifically focused on TBI, are crucial in assessing the safety and efficacy of new treatments. These trials serve as fundamental instruments in determining whether emerging medications outperform standard therapies, providing compelling evidence to support wider implementation.

The main goal is to thoroughly scrutinize trial completion rates and voluntary withdrawals among this particular group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document
* Participant must be 18 years of age or older
* Confirmed diagnosis of TBI

Exclusion Criteria:

* Enrolled in another research study
* Is pregnant, breastfeeding or expecting to conceive within the projected duration of the study
* Inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with TBI who are actively considering enrolling in a clinical study for said condition, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of TBI patients who decide to enroll in a clinical research | 3 months
Rate of TBI patients who remain in clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Perry DC, Sturm VE, Peterson MJ, Pieper CF, Bullock T, Boeve BF, Miller BL, Guskiewicz KM, Berger MS, Kramer JH, Welsh-Bohmer KA. Association of traumatic brain injury with subsequent neurological and psychiatric disease: a meta-analysis. J Neurosurg. 2016 Feb;124(2):511-26. doi: 10.3171/2015.2.JNS14503. Epub 2015 Aug 28. PMID 26315003
- [Background] Kaur P, Sharma S. Recent Advances in Pathophysiology of Traumatic Brain Injury. Curr Neuropharmacol. 2018;16(8):1224-1238. doi: 10.2174/1570159X15666170613083606. PMID 28606040
- [Background] VanderVeen JD. TBI as a Risk Factor for Substance Use Behaviors: A Meta-analysis. Arch Phys Med Rehabil. 2021 Jun;102(6):1198-1209. doi: 10.1016/j.apmr.2020.10.112. Epub 2020 Nov 2. PMID 33152264

DOCUMENTS (1):
  • Informed Consent Form (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT06288698/ICF_000.pdf